CLINICAL TRIAL: NCT01189370
Title: A Phase II Study of the Efficacy and Tolerability of the Dose Escalation of Sorafenib in Advanced Renal Cell Cancer
Brief Title: Evaluate Safety and Tolerability in Dose Escalation of Sorafenib in Advanced Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11277
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Cancer
Keywords: carcinoma, renal cell; kidney; cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-Patient Dose Escalation: Sorafenib (Experimental): All patients will receive a starting dose of sorafenib 400 mg by mouth twice daily. At four weeks, all patients who have not experienced Grade 3 or 4 toxicity will undergo dose escalation using a treatment schedule of days 1-5 days of each week. Doses will continue to be escalated every 4 weeks depending on tolerability and tumor response.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — Dose Level:
  1. 400mg twice daily, continuous.
  2. 600mg twice daily, days 1-5 of each week.
  3. 800mg twice daily, days 1-5 of each week.
  Other Names: BAY 43-9006; Nexavar®

SUMMARY:
The purpose of this study is to determine whether an increase in the dose of sorafenib when given over five instead of 7 days/week, will result in an improvement of the response rate (degree of shrinkage of your cancer) and an improvement in the length of time that sorafenib will control your cancer, without causing a significant increase in side effects.

DETAILED DESCRIPTION:
In 2006, an estimated 38,890 people in the United States were diagnosed with kidney cancer and greater than 12,000 died from the disease. Kidney cancer that has spread to other parts of the body is one of the most treatment-resistant diseases. Standard of care treatment usually involves chemotherapy. Results from chemotherapy have been disappointing. Therefore, there is a need to develop additional safe and effective therapies to treat advanced kidney cancer.

Sorafenib (Nexavar®) has been approved by the FDA for the treatment of advanced kidney cancer. Sorafenib works by interfering with a type of protein in your body that determines how your kidney cells work and grow. Sorafenib at standard doses for 400mg(two pills) twice/day, given seven days/week, may slow progression of the disease for an average of three months but it is not expected to be curative. Preliminary studies have suggested higher doses of sorafenib may increase the chance that the tumor will shrink.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0 grams per deciliter (g/dl)
  * Absolute neutrophil count (ANC)≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * and aspartate aminotransferase (AST) ≤ 2.5 times the ULN (≤ 5 x ULN for patients with liver involvement)
  * Creatinine < 1.5 times ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and willing to sign written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* International normalized ratio (INR) < 1.5 or a prothrombin time/partial prothrombin time (PT/PTT) within normal limits unless receiving anti-coagulation treatment with an agent such as warfarin or heparin. These patients may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Must have histologically or cytologically confirmed renal cell carcinoma that is metastatic (M1). Patients with unresectable primary tumor (but MO) are also eligible.
* Must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension. Soft tissue disease that has been radiated in the 2 months prior to registration is not assessable as measurable disease. Soft tissue disease within a prior radiation field must have progressed to be considered assessable. X-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration. X-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration.
* Patients with metastatic disease who have a resectable primary tumor and are deemed a surgical candidate may have undergone resection and have recovered from surgery. At least 28 days must have elapsed since surgery and must have recovered from any adverse effects of surgery.
* May have received 1 prior immunotherapy with either interferon (IFN) and/or Interleukin-2 (IL-2) or the combination of IFN/IL2 and only 1 prior biologic agent (sunitinib, bevacizumab, or temsorlimus). Must have progressed during this prior therapy. At least 14 days must have elapsed since the last treatment and must have recovered from any adverse effects of prior therapy. May have received prior radiation therapy. At least 21 days must have elapsed since completion of prior radiation therapy. Must have recovered from all associated toxicities at the time of registration.

Exclusion Criteria

* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Patients who have received prior sorafenib are ineligible.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B/C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombosis or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months. Patients with renal or caval thrombosis related to the primary renal tumor would not be excluded and are eligible.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Williamson, MD, Study Chair — The University of Kansas - Cancer Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 400mg: Participants were administered 400 mg of Sorafenib by mouth twice daily for 4 weeks, and were evaluated at four weeks for toxicity. At four weeks, all participants who have not experienced Grade 3 or 4 toxicity will undergo dose escalation.
- Cohort 2: 600 mg: Participants were administered 600mg of Sorafenib by mouth twice daily, days 1-5 of each week for 4 weeks, and were evaluated at four weeks for toxicity. At four weeks, all participants who have not experienced Grade 3 or 4 toxicity will undergo dose escalation.
- Cohort 3: 800mg: Participants were administered 800mg of Sorafenib by mouth twice daily, days 1-5 of each week for 4 weeks, and were evaluated at four weeks for toxicity. At four weeks, all participants who have not experienced Grade 3 or 4 toxicity will undergo dose escalation.
Period: Dose Level 1
Arm/Group | Cohort 1: 400mg | Cohort 2: 600 mg | Cohort 3: 800mg
Started | 25 | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 9 | 0 | 0
Period: Dose Level 2
Arm/Group | Cohort 1: 400mg | Cohort 2: 600 mg | Cohort 3: 800mg
Started | 0 | 16 | 0
Completed | 0 | 12 | 0
Not Completed | 0 | 4 | 0
Period: Dose Level 3
Arm/Group | Cohort 1: 400mg | Cohort 2: 600 mg | Cohort 3: 800mg
Started | 0 | 0 | 12
Completed | 0 | 0 | 6
Not Completed | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib: * Sorafenib 400 mg twice daily, 7 days a week
  * Sorafenib 600 mg twice daily, days 1-5 per week
  * Sorafenib 800 mg twice daily, days 1-5 per week
  * Sorafenib 1000 mg twice daily, says 1-5 per week
Arm/Group | Sorafenib
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Could Tolerate Each Dose Level
Description: Tolerability will be defined as successful completion of the dose level without experiencing Grade 3 or 4 toxicity.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 400mg | Cohort 2: 600 mg | Cohort 3: 800mg
Number analyzed (Participants) | 25 | 16 | 12
Participants
  Started Dose Level | 25 | 16 | 12
  Completed Dose Level | 16 | 12 | 6

2. Secondary Outcome: Overall Number of Participants That Had Disease Progression on Study
Description: Disease Progression as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Time Frame: 26 months
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Disease Progression: Total number of participants that had disease progression while on study. Disease progression based on RECIST criteria.
Arm/Group | Number of Participants With Disease Progression
Number analyzed (Participants) | 25
Participants | 17

ADVERSE EVENTS:
Groups:
- Sorafenib: * Sorafenib 400 mg twice daily, 7 days a week
  * Sorafenib 600 mg twice daily, days 1-5 per week
  * Sorafenib 800 mg twice daily, days 1-5 per week
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 14/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Intra-operative injury - Joint (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Pain (General disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Treatment related secondary malignancy (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=25)
Abdominal distention (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (9)
Acne (Skin and subcutaneous tissue disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)
Anorexia (Gastrointestinal disorders) | 14 (23)
Anxiety (Psychiatric disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Chest pain (Cardiac disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 13 (14)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
decubitus (Skin and subcutaneous tissue disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 18 (39)
Dizziness (Nervous system disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Ear, nose and throat examination abnormal (Ear and labyrinth disorders) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 5 (8)
Edema: head and neck (Blood and lymphatic system disorders) | 2 (2)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Esophogeal mucositis (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Pain: external ear (Ear and labyrinth disorders) | 1 (1)
fatigue (General disorders) | 19 (33)
fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 3 (4)
fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hand and foot syndrome (Infections and infestations) | 15 (31)
headache (Nervous system disorders) | 3 (4)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (12)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 3 (5)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (6)
joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (10)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (7)
Musculoskeletal - Other (Specify) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (22)
Neutrophils (Blood and lymphatic system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 5 (5)
Otitis, external (Ear and labyrinth disorders) | 1 (1)
Pain - Other (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11)
Pain: skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: pelvic (Reproductive system and breast disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 2 (3)
Platelets (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (5)
Psychosis (Psychiatric disorders) | 1 (1)
Pulmonary - Other(specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (16)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Pain: scalp (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Speech impairment (Nervous system disorders) | 1 (1)
Pain: stomach (Gastrointestinal disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 3 (4)
Taste alteration (Gastrointestinal disorders) | 6 (8)
Thrombosis (Vascular disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vaginitis (Reproductive system and breast disorders) | 1 (1)
Valvular heart disease (Cardiac disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (12)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes